CLINICAL TRIAL: NCT03023475
Title: Prospective Randomized Comparison of Two Different Endoscopic Radial Artery Harvesting Devices
Brief Title: Comparison of Two Different Endoscopic Radial Artery Harvesting Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerckhoff Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VesselHarvestingLigaSure
Record Dates: First submitted 2017-01-08; First posted 2017-01-18 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: CABG Graft Integrity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LigaSure endoscopic radial harvesting (Active Comparator): The endoscopic vessel harvesting will be performed using the LigaSure device.
  Interventions: Device: LigaSure endoscopic vessel harvesting
- TLS2 endoscopic radial harvesting (Active Comparator): The endoscopic vessel harvesting will be performed using the TLS2 device.
  Interventions: Device: TLS2 endoscopic vessel harvesting

INTERVENTIONS:
Device: LigaSure endoscopic vessel harvesting — The radial artery will be harvested endoscopically using the LigaSure system.
  Arms: LigaSure endoscopic radial harvesting
Device: TLS2 endoscopic vessel harvesting — The radial artery will be harvested endoscopically using the TLS2 system.
  Arms: TLS2 endoscopic radial harvesting

SUMMARY:
Endoscopic radial artery harvesting in coronary bypass surgery is routinely performed by the investigators. In this study, the investigators want to compare the MiFusion TLS2 (Endotrust GmbH, Germany) device to the LigaSure Maryland Jaw (Medtronic, USA). The vessel harvesting is performed in the standard fashion according to the institutional routine. The patients are randomized preoperatively to one of the devices. The proximal end of the radial artery will be preserved and deep-frozen for histological assessment. Endothelial integrity will be investigated using Hematoxylin-Eosin, CD31 and endothelial nitrogen monoxide synthase.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients undergoing CABG using the radial artery
* capability to give informed consent

Exclusion Criteria:

* no specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Endothelial integrity of the radial artery using histological examination. | Through study completion, an average of 1 year.

SECONDARY OUTCOMES:
Harvesting time | The harvesting time will be measured during the vessel harvesting surgery.
Hemostasis in the arm indicated by bleeding from radial artery side branches or veins in the arm. | Intraoperatively and directly after vessel harvesting the arm is controlled using the endoscope and bleeding can be detected during this control. End of surgery is end of this outcome parameter.
Accuracy of vessel sealing, if side branches of the radial artery are bleeding after blood insufflation, additional clips have to placed at the side branch. | The blood insufflation is performed immediately after vessel harvesting and leaks can be detected.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Van Linden, MD, Principal Investigator — Kerckhoff Klinik
Locations (1):
- Kerckhoff Klinik, Bad Nauheim, Germany

IPD SHARING:
Plan to Share IPD: No